CLINICAL TRIAL: NCT05709184
Title: Lyophilized Fecal Microbiome Transfer for Primary Clostridioides Difficile Infection (DONATE Study): a Multicenter Randomized Controlled Trial
Brief Title: Lyophilized Fecal Microbiome Transfer vs. Vancomycin Monotherapy for Primary Clostridioides Difficile Infection
Acronym: DONATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); European Institute of Oncology (Other); University of Alberta (Other); Imperial College London (Other); University of Debrecen (Other); Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Milena Pitashny, MD, Director of Clinical and Research Microbiome Center, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMB-0176-22
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Clostridioides Difficile Infection
Keywords: Gut microbiome; Colonization resistance; Fecal microbiome transfer; Lyophilization; Multi-drug resistant organisms; Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome will be assessed by an observer blinded to study group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lyophilized fecal microbiome transfer (Lyo-FMT) (Experimental): Vancomycin will be given orally in 125 mg capsules/solution 4 times daily for a total of 5 days (day 1 - initiation of therapy by the clinical team), followed by a loading dose of oral Lyo-FMT capsules on day 6 (15 capsules). On days 7-10, patients will receive 10 Lyo-FMT capsules per day. A total of 55 capsules, derived from ~30-40g of the original material, will be administered throughout 5 days. Prior to each Lyo-FMT administration, patients will be asked to fast for 8 hours. Bowel preparation or proton pump inhibitor use will not be required per protocol. The loading dose will be administered under medical supervision, while further dosing can be administered at the patient's home/institute, after training and guidance
  Interventions: Combination Product: Lyophilized fecal microbiome transfer
- Vancomycin monotherapy (Active Comparator): Vancomycin will be given orally in 125 mg capsules/solution 4 times daily for a total of 10 days (day 1 - initiation of therapy by the clinical team, not from randomization).
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Combination Product: Lyophilized fecal microbiome transfer — Five days of vancomycin followed by five days of lyophilized fecal microbiome transfer, administered in a loading dose of 15 capsules, and a daily maintenance dose of 10 capsules.
  Other Names: FMT
  Arms: Lyophilized fecal microbiome transfer (Lyo-FMT)
Drug: Vancomycin — Ten days of oral vancomycin 125 mg four times daily
  Other Names: CDI antibiotic treatment
  Arms: Vancomycin monotherapy

SUMMARY:
The goal of this clinical trial is to test whether lyophilized fecal microbime transfer - a dried extract of bacteria from the stool of healthy donors - is better than antibiotic therapy only for treating primary clostridioides difficile infection (CDI) in adult participants.

The main question it aims to answer is whether lyophilized fecal microbiome transfer lowers the number of episodes of CDI compared to antibiotic therapy.

Participants will be assigned to one of two groups:

* In the intervention group participants will be given vancomycin by mouth for five days followed by 5 days of capsules of lyophilized fecal microbiome to swallow, up until day 10.
* In the control group participants will be given vancomycin by mouth for ten days.
* All participants will be asked to arrive for two follow-up visits and to fill out questionnaires. In addition, all participants will be asked to give stool samples before antibiotic therapy and on the two follow-up visits.

Researchers will compare the intervention group and the control group to see if there is a difference in symptoms degree after ten days and in recurrence of the infection after two months. They will also compare side effects, the total use of antibiotics and the change in the composition of bacteria in the stool, namely the presence of bacteria that are resistant to many drugs.

DETAILED DESCRIPTION:
This is a multicenter, transnational randomized controlled trial comparing a short course of vancomycin therapy followed by oral lyophilized fecal microbiome transfer (Lyo-FMT) capsules (intervention group) with standard vancomycin monotherapy (control group), for adults with primary Clostridioides difficile infection (pCDI).

The target population will be adult patients with non-fulminant pCDI in the community/hospital according to the setting at the recruiting center. pCDI will be defined as the patient's first event of CDI in the last 6 months presenting with a new-onset diarrhea (≥3 unformed bowel movements per day for more than 24 hours) and laboratory detection of toxigenic C. difficile in feces. A positive C. difficile stool sample will be defined per study center according to international guidelines, with an obligatory positive toxin test to assure the presence of an active toxigenic CD strain. Both non-severe and severe patients will be included.

Consenting patients will be randomly assigned to one of two treatment modalities: vancomycin followed by oral lyophilized FMT capsules (intervention group) or vancomycin monotherapy group.

* Lyo-FMT group (intervention group) - vancomycin will be given orally in 125 mg capsules/solution 4 times daily for a total of 5 days (day 1 - initiation of antibiotic therapy by the clinical team), followed by a loading dose of oral lyophilized FMT capsules on day 6 (15 capsules). On days 7-10, patients will receive 10 Lyo-FMT capsules per day. A total of 55 capsules, derived from ~30-40g of the original material, will be administered throughout 5 days. Prior to each FMT administration, patients will be asked to fast for 8 hours. Bowel preparation or proton pump inhibitor use will not be required per protocol. The loading dose will be administered under medical supervision, while further dosing can be administered at the patient's home/institute, after training and guidance.
* Antibiotic monotherapy group (control group) - vancomycin will be given orally in 125 mg capsules/solution 4 times daily for a total of 10 days (day 1 - initiation of therapy by the clinical team, not from randomization).

If symptoms persist on day 10 from the initiation of therapy, further treatment will be given according to study group allocation. In the Lyo-FMT group, FMT will be repeated in the form of 15 FMT capsules per course as clinically indicated. If no resolution of symptoms will be documented after 2 days of FMT, the same FMT course (15 capsules) will be repeated, up to 3 times. For patients in the antibiotic monotherapy group, an extension of the vancomycin treatment with the same doses will be given for 7 more days. Laboratory testing for the presence of C. difficile will not be required for the administration of repeated treatment, but will be annotated if performed. If symptoms will persist beyond day 18 of the study in both groups (8 days after the end of first treatment), we will allow treatment according to clinical judgement at the local study center. Patients will be free to decide if they want to stop their participation in the study at all times. Persistent symptoms beyond day 20 of the study will be considered as a clinical failure for the purposes of secondary outcome analysis. At any point, if there is a deterioration of the patient towards fulminant disease, clinical judgement will prevail as per protocol for fulminant cases.

During the study period and across study centers, we will encourage clinicians to use vancomycin as empiric treatment for pCDI. However, according to local clinical practice, patients may receive an antibiotic other than vancomycin (e.g. metronidazole). In both study groups, patients that were treated with another antibiotic agent in the first 24 hours, will be switched to vancomycin prior to day 3 of the study. The day of initiation of therapy will be considered from the first day of any antibiotic therapy that was administered. Randomization will be done within 72 hours from the initiation of any therapy for CDI.

In both groups, if a patient receives concurrent systemic antibiotics for other indications, the research team will contact the clinical team to understand if these antibiotics can be safely stopped 24 hours prior to randomization (day 3 from initiation of therapy). If systemic antibiotics cannot be stopped, then the patient will be excluded from the study.

In case of a CDI recurrence, the patient will be considered as reaching the primary outcome. We will permit treatment of CDI recurrences according to clinical judgement. We will provide Lyo-FMT for the treatment of recurrent CDI If available at the study center and required by the clinical team. In case of the development of fulminant disease, we will allow any therapy judged by the clinical team as appropriate. All cases with fulminant disease will be assessed by a surgical team for a timely fashioned colectomy if indicated. The development of fulminant disease from day 8 of the study onwards (3 days on FMT treatment) will be considered as clinical failure for the purposes of secondary outcome analysis.

The trial's primary efficacy outcome is the recurrence of CDI by week 8. Recurrence will be defined as the re-appearance of CDI symptoms (at least 3 unformed bowel movements per day for at least 2 days) with positive C. difficile stool test more than 3 days after the resolution of symptoms and requiring anti-CDI treatment. The primary outcome will be assessed by an observer blinded to study group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults ≥18 years old with non-fulminant primary CDI.
* Both non-severe and severe patients will be included.
* Primary CDI (pCDI) will be defined as the patient's first event of CDI in the past 6 months: New-onset diarrhea (≥3 unformed bowel movements (UBM) per day for more than 24 hours) and laboratory detection of toxigenic C. difficile in feces.
* A positive CD stool sample will be defined per study center according to international guidelines, with an obligatory positive toxin test to assure the presence of an active toxigenic CD strain.

Exclusion Criteria:

* Patients who cannot provide informed consent and do not have a legal guardian;
* History of CDI 6 months prior to screening
* Known presence of other stool pathogens known to cause diarrhea;
* Patients who cannot swallow;
* Background diagnosis of inflammatory bowel disease, irritable bowel syndrome (IBS), or any other chronic diarrheal disorder;
* Active gastrointestinal graft versus host disease (GVHD);
* Neutropenia <500/ml3;
* Food allergy leading to anaphylaxis;
* Prior total colectomy or the presence of a small intestinal stoma;
* Perforated intestine or intestinal fistula or major abdominal surgery in the last 30 days;
* Fulminant or life-threatening CDI defined as the occurrence of ileus, septic shock or toxic megacolon. Signs of fulminant disease are: white blood cell count >30,000 cells/mL; temperature >40°C; evidence of hypotension [systolic blood pressure <90 mmHg], peritoneal signs, and significant dehydration;
* Early fulminant CDI (ICU patients) defined as patients showing progression despite treatment with a sequential organ failure assessment score (SOFA score) ≥ 4 due to CDI (13) at day 2 of treatment (prior to randomization);
* Patients who receive systemic antibiotics due to other reasons which cannot be stopped until 1 day prior to randomization (day 2 of antibiotic therapy);
* Patients that were not recruited to the study by day 4 of CDI therapy will be excluded from participation;
* Patients with <3 months life expectancy;
* Inability or unwillingness to comply with the study protocol, including ingesting capsules, and providing blood or stool samples as scheduled;
* Participation in another interventional study;
* In the opinion of the investigator, inappropriateness for the trial (eg, patients with known hypersensitivity to vancomycin);
* Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
CDI recurrence | 8 weeks
  The re-appearance of CDI symptoms (at least 3 unformed bowel movements per day for at least 2 days) with positive CD stool test more than 3 days after the resolution of symptoms and requiring anti-CDI treatment

SECONDARY OUTCOMES:
Clinical cure | 10 days
  Cessation of CDI related symptoms by day 10 of the study with no further symptoms/conditions (persistent symptoms, fulminant disease, death and colectomy) needing additional therapy
CDI recurrence in patients who achieved clinical cure | 8 weeks
  CDI recurrence in patients who achieved clinical cure at day 10
Sustained clinical response | 8 weeks
  Cessation of CDI related symptoms by day 10 of the study with no further symptoms/conditions (persistent symptoms, fulminant disease, death, colectomy and recurrence) needing additional therapy
Serious adverse events | 8 weeks
  Mortality, bacteremia attributable to FMT, and hospitalization due to CDI during study period
Patient reported outcomes (PROs) and preferences | At baseline and 8 weeks
  The C. difficile health-related quality of life (HRQOL) questionnaire,13 EuroQol 5 Dimensions 5 Level (EQ-5D-5L),14 and Work Productivity and Activity Impairment (WPAI) Questionnaire15 will be administered at screening visit and again at week 2, and week 8. The C difficile HRQOL questionnaire is specifically developed and validated to assess patients with CDI. Although EQ-5D-5L and WPAI are not specifically designed for patients with CDI, they are well validated instruments and have been used in clinical research across a variety of conditions and health status. If follow-up visits are deemed non-essential and are conducted by phone, these questionnaires may be emailed out or mailed out to patients based on patient preference and to be returned to the study sites.
Patient preference for treatment | At baseline and week 8
  A patient preference questionnaire designed by the investigators

OTHER OUTCOMES:
Time to clinical cure | up to 10 days
  Days until clinical cure from day 1
Time to recurrence | up to 8 weeks
  Days until recurrence from reported clinical cure
Total adverse events rate | 8 weeks
  The rate of all adverse events during the trial.
Acquisition of multidrug-resistant organisms carriage | 8 weeks
  Acquisition of carbapenem-resistant Enterobacterales, vancomycin-resistant Enterococcus and Extended Spectrum Beta-Lactamase producing Enterobacterales
Changes in intestinal resistome | 14 days and 8 weeks
  Changes in antibiotic resistance genes and bacteria
Shifts in the microbial community | 14 days and 8 weeks
  Changes in gut microbiome

CONTACTS AND LOCATIONS:
Locations (6):
- University of Alberta, Edmonton, Canada
- University of Debrecen, Debrecen, Hungary
- Rambam Health Care Campus, Haifa, Israel
- Gemelly institute Policlinico Universitario Fondazione Agostino Gemelli, Rome, Italy
- Hospital of Lithuania University of Health Sciences Kauno klinikos, Kaunas, Lithuania
- Imperial College of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawson PA, Citron DM, Tyrrell KL, Finegold SM. Reclassification of Clostridium difficile as Clostridioides difficile (Hall and O'Toole 1935) Prevot 1938. Anaerobe. 2016 Aug;40:95-9. doi: 10.1016/j.anaerobe.2016.06.008. Epub 2016 Jun 28. PMID 27370902
- [Background] Lessa FC, Mu Y, Bamberg WM, Beldavs ZG, Dumyati GK, Dunn JR, Farley MM, Holzbauer SM, Meek JI, Phipps EC, Wilson LE, Winston LG, Cohen JA, Limbago BM, Fridkin SK, Gerding DN, McDonald LC. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Feb 26;372(9):825-34. doi: 10.1056/NEJMoa1408913. PMID 25714160
- [Background] Lewis BB, Buffie CG, Carter RA, Leiner I, Toussaint NC, Miller LC, Gobourne A, Ling L, Pamer EG. Loss of Microbiota-Mediated Colonization Resistance to Clostridium difficile Infection With Oral Vancomycin Compared With Metronidazole. J Infect Dis. 2015 Nov 15;212(10):1656-65. doi: 10.1093/infdis/jiv256. Epub 2015 Apr 28. PMID 25920320
- [Background] Rewers M, Hyoty H, Lernmark A, Hagopian W, She JX, Schatz D, Ziegler AG, Toppari J, Akolkar B, Krischer J; TEDDY Study Group. The Environmental Determinants of Diabetes in the Young (TEDDY) Study: 2018 Update. Curr Diab Rep. 2018 Oct 23;18(12):136. doi: 10.1007/s11892-018-1113-2. PMID 30353256
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Adler A, Miller-Roll T, Bradenstein R, Block C, Mendelson B, Parizade M, Paitan Y, Schwartz D, Peled N, Carmeli Y, Schwaber MJ. A national survey of the molecular epidemiology of Clostridium difficile in Israel: the dissemination of the ribotype 027 strain with reduced susceptibility to vancomycin and metronidazole. Diagn Microbiol Infect Dis. 2015 Sep;83(1):21-4. doi: 10.1016/j.diagmicrobio.2015.05.015. Epub 2015 Jun 3. PMID 26116225
- [Background] Huttner BD, de Lastours V, Wassenberg M, Maharshak N, Mauris A, Galperine T, Zanichelli V, Kapel N, Bellanger A, Olearo F, Duval X, Armand-Lefevre L, Carmeli Y, Bonten M, Fantin B, Harbarth S; R-Gnosis WP3 study group. A 5-day course of oral antibiotics followed by faecal transplantation to eradicate carriage of multidrug-resistant Enterobacteriaceae: a randomized clinical trial. Clin Microbiol Infect. 2019 Jul;25(7):830-838. doi: 10.1016/j.cmi.2018.12.009. Epub 2019 Jan 4. PMID 30616014
- [Background] Juul FE, Garborg K, Bretthauer M, Skudal H, Oines MN, Wiig H, Rose O, Seip B, Lamont JT, Midtvedt T, Valeur J, Kalager M, Holme O, Helsingen L, Loberg M, Adami HO. Fecal Microbiota Transplantation for Primary Clostridium difficile Infection. N Engl J Med. 2018 Jun 28;378(26):2535-2536. doi: 10.1056/NEJMc1803103. Epub 2018 Jun 2. No abstract available. PMID 29860912
- [Background] Camacho-Ortiz A, Gutierrez-Delgado EM, Garcia-Mazcorro JF, Mendoza-Olazaran S, Martinez-Melendez A, Palau-Davila L, Baines SD, Maldonado-Garza H, Garza-Gonzalez E. Randomized clinical trial to evaluate the effect of fecal microbiota transplant for initial Clostridium difficile infection in intestinal microbiome. PLoS One. 2017 Dec 20;12(12):e0189768. doi: 10.1371/journal.pone.0189768. eCollection 2017. PMID 29261736
- [Background] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- [Background] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878
- [Background] Staley C, Hamilton MJ, Vaughn BP, Graiziger CT, Newman KM, Kabage AJ, Sadowsky MJ, Khoruts A. Successful Resolution of Recurrent Clostridium difficile Infection using Freeze-Dried, Encapsulated Fecal Microbiota; Pragmatic Cohort Study. Am J Gastroenterol. 2017 Jun;112(6):940-947. doi: 10.1038/ajg.2017.6. Epub 2017 Feb 14. PMID 28195180
- [Background] Reigadas E, Bouza E, Olmedo M, Vazquez-Cuesta S, Villar-Gomara L, Alcala L, Marin M, Rodriguez-Fernandez S, Valerio M, Munoz P. Faecal microbiota transplantation for recurrent Clostridioides difficile infection: experience with lyophilized oral capsules. J Hosp Infect. 2020 Jun;105(2):319-324. doi: 10.1016/j.jhin.2019.12.022. Epub 2019 Dec 26. PMID 31883938
- [Background] Haifer C, Paramsothy S, Borody TJ, Clancy A, Leong RW, Kaakoush NO. Long-Term Bacterial and Fungal Dynamics following Oral Lyophilized Fecal Microbiota Transplantation in Clostridioides difficile Infection. mSystems. 2021 Feb 2;6(1):e00905-20. doi: 10.1128/mSystems.00905-20. PMID 33531405